CLINICAL TRIAL: NCT02206646
Title: Post Marketing Surveillance to Monitor the Safety and Efficacy of Metalyse® (Tenecteplase) in Korean Patients With Acute Myocardial Infarction
Brief Title: Post Marketing Surveillance to Monitor the Safety and Efficacy of Metalyse® in Korean Patients With Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1123.25
Record Dates: First submitted 2014-07-31; First posted 2014-08-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Tenecteplase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Metalyse: weight-adjusted dose
  Interventions: Drug: Metalyse

INTERVENTIONS:
Drug: Metalyse

SUMMARY:
To monitor the safety of Metalyse® in clinical practice in patients with acute myocardial infarction over a period of 6 years as required by Korean authorities, with the following observations:

1. Unexpected adverse drug reactions
2. Frequency and nature of adverse events (AEs)
3. Factors on the safety and efficacy profile of the Metalyse® Injection. Efficacy of Metalyse® was also assessed.

ELIGIBILITY:
Inclusion Criteria:

* none

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed with acute myocardial infarction
Sampling Method: Non-Probability Sample
Enrollment: 987 (Actual)
Dates: Start 2003-02; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
30-day mortality after the Metalyse® Injection | 30 days
Outcome assessment - 'Improvement' or 'Failure' | 30 days
  'Improvement' was defined as survival on 30 days and 'Failure' as death on 30 days after the Metalyse treatment.
Number of patients with adverse events | up to 30 days